CLINICAL TRIAL: NCT03279822
Title: Association Analysis for Chronic Diseases Based on Resident Health Records in China by Using Big Data Methods
Brief Title: Association Analysis for Chronic Diseases Based on Resident Health Records by Using Big Data Methods
Status: Completed | Type: Observational
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zihui Tang, Principal Investigator, Huashan Hospital
Other Study IDs: 20170905
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group
  Interventions: Other: not any intervention

INTERVENTIONS:
Other: not any intervention — not any intervention

SUMMARY:
This is an observational study to analysis the association factors for common diseases, including chronic obstructive pulmonary disease, coronary artery disease, hypertension, diabetes etc, based on resident healthcare records. More than 10 million resident healthcare records should be collected for the associations study by using big data methods.

ELIGIBILITY:
Inclusion Criteria:

* Survey Chinese residents aged 20 - 100 years, were included in this study.

Exclusion Criteria:

* Serious hepatic or renal dysfunctions.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators collect data regarding residents health records from rural and urban in China. This study needs more than 10 million resident records from 2010.
Sampling Method: Non-Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
regular diagnosis and medical history of common diseases | an average of 1 year
  resident health records for medical history of common diseases, questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Huasha Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu J, Xu F, Mohammadtursun N, Lv Y, Tang Z, Dong J. The Analysis of Constitutions of Traditional Chinese Medicine in Relation to Cerebral Infarction in a Chinese Sample. J Altern Complement Med. 2018 May;24(5):458-462. doi: 10.1089/acm.2017.0027. Epub 2017 Aug 18. PMID 28820606
- [Background] Li X, Lei T, Tang Z, Dong J. Analyzing the association between fish consumption and osteoporosis in a sample of Chinese men. J Health Popul Nutr. 2017 Apr 19;36(1):13. doi: 10.1186/s41043-017-0088-y. PMID 28424092